CLINICAL TRIAL: NCT05428059
Title: The Effect of Mobile Health-Education Application on Healthy Lifestyle Behaviors in Patients Planned for Bariatric Surgery:A Randomized Controlled Study
Brief Title: The Effect of Mobile Health-Education Application on Healthy Lifestyle Behaviors in Patients Planned for Bariatric Surgery
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was interrupted due to the small number of patients constituting the sample.
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Sevgi Deniz Dogan, lecturer Dr., Cukurova University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 5312256943
Record Dates: First submitted 2022-06-15; First posted 2022-06-22 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Nursing Caries; Bariatric Surgery Candidate; Mobile Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- application group (Experimental): In addition to standard care, training and consultancy will be provided with a mobile application.
  Interventions: Other: mobile education
- control group (No Intervention): Standard care will be given

INTERVENTIONS:
Other: mobile education — The training content prepared by the researchers will be presented to the expert opinion. After the necessary arrangements, it will be installed on the mobile application. The mobile application will be downloaded to the patients' phones for one month. It will be in live consultation.
  Arms: application group

SUMMARY:
Obesity, which is the second leading cause of preventable death in the world, affects all the systems in the body and affects many physiological problems, as well as the mental state, body image and quality of life of the individual. For this reason, obese individuals try various treatment methods in order to get rid of obesity, and in cases where these methods fail, they often prefer bariatric surgery. It is very important that patients who will undergo bariatric surgery can adapt to the anatomical changes in their body and shape their lifestyle accordingly. Otherwise, it is inevitable for patients to face various complications after surgery. After bariatric surgery, a structured training program in the preoperative period is of great importance in order for the patient to adapt to the changes in his body, to prevent the development of possible complications, to be affected by the negativities that may occur due to the current change, and to prepare for the new lifestyle. In this context, the main subject of this research is to enable individuals to gain healthy lifestyle behaviors by providing mobile-based training and consultancy services that enable them to easily access the right information at the desired time and place.

ELIGIBILITY:
Inclusion Criteria:

* Being literate,
* Being able to understand, speak Turkish and not have a hearing impairment,
* First time to undergo bariatric surgery,
* Absence of any psychiatric disorder that will reduce the ability to comprehend and understand,
* Ability to use Android-based smartphones,
* Agreeing to participate in the research.

Exclusion Criteria:

* Patient's desire to quit the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
The Effect of Mobile Health-Education Application on Healthy Lifestyle Behaviors in Patients Planned for Bariatric Surgery | one months
  Data will be evaluated using the Healthy Lifestyle Behaviors Scale-II. The minimum score that can be obtained from the 52-item scale is 52, and the maximum score is 208. A high score from the scale indicates that individuals have good HLPS levels, and low scores indicate bad HLBD.

CONTACTS AND LOCATIONS:
Locations (1):
- Çukurova University Institute of Health Sciences, Adana, Turkey (Türkiye)